CLINICAL TRIAL: NCT07362537
Title: Enteral Nutrition Delivery in Prone Position Ventilated Patients With Moderate to Severe Acute Respiratory Distress Syndrome: a Randomized Controlled Trial
Brief Title: Enteral Nutrition Delivery in Prone Position Ventilated Patients With Moderate to Severe ARDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Professor, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20231030 prone nutrition
Record Dates: First submitted 2024-04-01; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: ARDS
Keywords: ARDS; prone position ventilation; enteral nutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-pyloric feeding group (Experimental): Enteral nutrition through nasojejunal tube
  Interventions: Procedure: enteral nutrition through nasojejunal tube
- Gastric feeding group (Active Comparator): Enteral nutrition through nasogastric tube
  Interventions: Procedure: enteral nutrition through nasogastric tube

INTERVENTIONS:
Procedure: enteral nutrition through nasojejunal tube — place nasojejunal tube for enteral nutrition
  Arms: Post-pyloric feeding group
Procedure: enteral nutrition through nasogastric tube — place nasogastric tube for enteral nutrition
  Arms: Gastric feeding group

SUMMARY:
This pilot study is aimed to compare and assess the impact, safety, and practical utility of gastric versus postpyloric feeding in moderate to severe ARDS patients with prone position ventilation. Patients included will be randomly assigned to receive enteral nutrition either through a nasogastric tube or a nasojejunal tube. The primary endpoint is the achievement of enteral nutrition goals. Secondary endpoints include the incidence of hospital-acquired infections, the number of ventilator-free days within 28 days, ICU length of stay, ICU mortality, 28-day mortality, 60-day mortality rates, the incidence of enteral nutrition intolerance, and the rate of enteral nutrition intake.

ELIGIBILITY:
Inclusion Criteria:

* ARDS patients who meet the Berlin criteria for ARDS and have a P/F ratio ≤ 200mmHg.
* Patients receiving invasive mechanical ventilation and clinically judged to require prone ventilation, with an anticipated daily prone positioning time of ≥12 hours and a duration of prone ventilation therapy of ≥3 days.
* Patients planned to receive enteral nutrition.
* Age ≥18 and ≤85 years.
* Consent to sign an informed consent form.

Exclusion Criteria:

* Contraindications to enteral nutrition, such as severe intestinal ischemia, active upper gastrointestinal bleeding, high-output intestinal fistula without a distal feeding route, abdominal compartment syndrome, severe diarrhea, intestinal obstruction, etc.
* Presence of shock with hemodynamic instability (norepinephrine or equivalent vasopressor dosage ≥0.5ug/kg.min) or tissue hypoperfusion (lactate >3mmol/L).
* Life-threatening hypoxemia, hypercapnia, and acidosis.
* Inability to tolerate prone ventilation (e.g., pregnant women, limb contractures, recent fractures, recent thoracic or abdominal surgery, pacemaker insertion within 48 hours, spinal instability, pelvic fractures, facial fractures, anticipated difficult airway).
* Conditions preventing nasogastric or nasojejunal tube placement (e.g., esophageal rupture, severe esophageal varices).
* Anticipated inability to start enteral nutrition within 48 hours.
* Use of prokinetic agents within 48 hours prior to starting enteral nutrition.
* Enteral nutrition via gastrostomy or jejunostomy.
* Expected ICU stay or survival time less than 3 days.
* Patients refusing further resuscitative treatment.
* Pregnant or breastfeeding women.
* Patients already enrolled in other interventional clinical studies or deemed unsuitable for the study by the clinician.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative Enteral Nutrition intake to target ratio | follow-up till 7-day
  The ratio of total calorie and protein intake through EN to target calorie and protein respectively.

SECONDARY OUTCOMES:
Incidence of new Infections | follow-up till 28-day
  New infections occur after admission to ICU within 28 days after admission to this study
Ventilator-free days within 28 days | follow-up till 28-day
  the number of days within a 28-day period that a patient does not require mechanical ventilation.
ICU Length of Stay | up to 24 weeks
  Duration of time a patient spends in the ICU from admission to discharge.
ICU Mortality Rate | up to 24 weeks
  The proportion of patients who die in the Intensive Care Unit (ICU) of a hospital
28-Day Mortality Rate | 28 days
  The proportion of patients who die within 28 days.
60-Day Mortality Rate | 60 days
  The proportion of patients who die within 60 days.
Incidence Rate of Enteral Nutrition Intolerance | 28 days
  The frequency at which patients experience intolerance to enteral feeding.
Daily Enteral Nutrition Intake Rate | 7 days
  It is calculated as the total volume of enteral nutrition fed to a patient each day, divided by the total prescribed enteral nutrition for that day, multiplied by 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda hospital, Southeast university, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
by email
Supporting Information: Study Protocol, SAP
Time Frame: Starting from the official publication of the manuscript to 1 year later
Access Criteria: collaborator